CLINICAL TRIAL: NCT06625801
Title: Intravascular Ultrasound Guidance for Complex High-risk Indicated Procedures in Underrepresented Patient Populations Registry
Brief Title: IVUS CHIP UPP Registry
Status: Not yet recruiting | Type: Observational
Sponsor: ECRI bv (Industry)
Collaborators: Boston Scientific Corporation (Industry); Cardialysis B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECRI-14-US
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease Risk High; Complex Coronary Artery Disease
Keywords: PCI; intravascular ultrasound; CHIP; ivus-guidance
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- IVUS-guided PCI in patients traditionally underrepresented in clinical trials: Patients undergoing IVUS-guided PCI for complex coronary artery disease who self-identify within a census-defined minority in the United States
  Interventions: Device: IVUS

INTERVENTIONS:
Device: IVUS — Intravascular Ultrasound

SUMMARY:
The IVUS CHIP UPP Registry is a prospective, observational, multicenter, single-arm registry. A total of 1010 patients with complex coronary lesions will be enrolled in up to 2 years, with at least 500 men and women. All patients will be treated with IVUS-guided PCI.

DETAILED DESCRIPTION:
Objective is to describe in a United States population the clinical efficacy and safety of an IVUS-guided approach in patients who self-identify within a census-defined minority undergoing PCI of complex coronary lesions, as well as clinical outcomes up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age and self-identify within a US census-defined minority
2. Patients with an indication for PCI of at least one lesion satisfying any of the following criteria:

   1. Angiographic heavy calcification
   2. Ostial lesions
   3. True bifurcation lesions involving side-branches >2.5mm
   4. Left main lesions
   5. Chronic total occlusion
   6. In-stent restenosis
   7. Long-lesions (estimated stent length > 28mm) OR Patient with an indication for PCI for any lesion and in need for elective mechanical circulatory support assisted PCI
3. Presenting with silent ischemia, stable angina, unstable angina or non-ST-elevation acute coronary syndrome (NSTE-ACS)
4. All lesions must be suitable for treatment with FDA-approved contemporary generation drug eluting stents or drug-coated balloons
5. The patient is willing and able to cooperate with registry procedures and follow-up until registry completion
6. Subject is able to confirm understanding of risks, benefits and treatment alternatives and he/she (or an authorized legal representative) provides informed consent prior to any protocol-related procedure, as approved by the appropriate IRB

Exclusion Criteria:

1. ST-elevation myocardial infarction or cardiogenic shock within prior 7 days
2. Known untreated severe valvular heart disease
3. Contraindication on the use of IVUS (i.e. extreme vessel tortuosity)
4. Requiring PCI in a diseased aorto-coronary bypass
5. Known contraindication or hypersensitivity to anticoagulants
6. Absolute contraindications or allergy that cannot be pre-medicated, to iodinated contrast or to antiplatelet drugs, including both aspirin and P2Y12 inhibitors
7. Non-cardiac co-morbidities with a life expectancy less than 1 year
8. A patients that is currently participating in a clinical trial that has not yet reached its primary endpoint cannot be included in this registry. A patient may only be enrolled in this registry once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients self-identified within a US census-defined minority with indication for IVUS-guided PCI of complex coronary lesions are consented for entering into the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Target-vessel failure (TVF) | 1 year after enrollment
  TVF is defined as a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target-vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Spitzer, MD, Study Director — European Cardiovascular Research Institute; David E Kandzari, MD, Principal Investigator — Piedmont Heart Institute

IPD SHARING:
Plan to Share IPD: No